CLINICAL TRIAL: NCT05898243
Title: Prospective Descriptive Study of Injuries Associated to Anterior Shoulder Dislocations in Patients Over 40 Years
Status: Recruiting | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Mònica Salomó Domènech, Doctor, Corporacion Parc Tauli
Other Study IDs: Dislocation
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Anterior Glenohumeral Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Humeral anterior dislocation: Patients presenting a first episode of humeral anterior dislocation and who are over 40 years old.
  Interventions: Procedure: Reduction

INTERVENTIONS:
Procedure: Reduction — An Rx will be performed before and after the reduction of the dislocation. After that, the neurovascular state will be checked and also if there is some associated injury.

SUMMARY:
The glenohumeral joint has the highest rate of dislocation of the whole body, due to its high mobility and the special characteristics of its anatomy. It is estimated that every year between 1-2% of the population will suffer from glenohumeral dislocation. The vast majority of studies are based on young patients under the age of 40, given that at this age they have the higher incidence and at the same time, they have higher redislocation index. However, the investigators are in front of a more active population with a longer life expectancy. That is why the cases of anterior glenohumeral dislocations are increasing in people older than 40 years. Given that most studies focus on younger patients, the investigators lack knowledge about which injuries are associated with dislocation at this age and whether these influence its clinical evolution.

ELIGIBILITY:
Inclusion Criteria:

* More than 40 years old
* First episode of traumatic anterior gelnohumeral dislocation seen in Rx
* Acceptance to be checked over 2 years
* Acceptance to be submitted to TAC, NMR, EMG and Bilateral Ultrasound

Exclusion Criteria:

* Previous fractures in this extremity
* Previous neurovascular lesions in this extremity
* Other associated lesions
* Cognitive alterations or dementia which prevent completing the protocols. Patients with <14 points in Mini-mental test.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with an anterior glenohumeral dislocation and over 40 years old who came to the Emergency Room in the Hospital between June 2023 and June 2025
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of associated lesions | At the three months visit including assessment of NMR/EMG/TAC/Bilateral Ultrasound

SECONDARY OUTCOMES:
Constant Functional Test | 3, 6, 12 and 24 months
WOSI test | 3, 6, 12 and 24 months
SST | 3, 6, 12 and 24 months
Redislocations | 3, 6, 12 and 24 months
Type of treatment | 3, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smartt AA, Wilbur RR, Song BM, Krych AJ, Okoroha K, Barlow JD, Camp CL. Natural History of First-Time Anterior Shoulder Dislocation in Patients Older Than 50 Years: A Study of 179 Patients With a Mean Follow-up of 11 Years. Orthop J Sports Med. 2022 Nov 2;10(11):23259671221129301. doi: 10.1177/23259671221129301. eCollection 2022 Nov. PMID 36339796
- [Background] Rapariz JM, Martin-Martin S, Pareja-Bezares A, Ortega-Klein J. Shoulder dislocation in patients older than 60 years of age. Int J Shoulder Surg. 2010 Oct;4(4):88-92. doi: 10.4103/0973-6042.79792. PMID 21655003
- [Background] Robinson CM, Shur N, Sharpe T, Ray A, Murray IR. Injuries associated with traumatic anterior glenohumeral dislocations. J Bone Joint Surg Am. 2012 Jan 4;94(1):18-26. doi: 10.2106/JBJS.J.01795. PMID 22218378
- [Background] Maier M, Geiger EV, Ilius C, Frank J, Marzi I. Midterm results after operatively stabilised shoulder dislocations in elderly patients. Int Orthop. 2009 Jun;33(3):719-23. doi: 10.1007/s00264-008-0578-z. Epub 2008 May 24. PMID 18500515
- [Background] Atef A, El-Tantawy A, Gad H, Hefeda M. Prevalence of associated injuries after anterior shoulder dislocation: a prospective study. Int Orthop. 2016 Mar;40(3):519-24. doi: 10.1007/s00264-015-2862-z. Epub 2015 Jul 2. PMID 26133290
- [Background] Sonnabend DH. Treatment of primary anterior shoulder dislocation in patients older than 40 years of age. Conservative versus operative. Clin Orthop Relat Res. 1994 Jul;(304):74-7. PMID 8020237
- [Background] Liavaag S, Stiris MG, Svenningsen S, Enger M, Pripp AH, Brox JI. Capsular lesions with glenohumeral ligament injuries in patients with primary shoulder dislocation: magnetic resonance imaging and magnetic resonance arthrography evaluation. Scand J Med Sci Sports. 2011 Dec;21(6):e291-7. doi: 10.1111/j.1600-0838.2010.01282.x. Epub 2011 Mar 15. PMID 21401723
- [Background] Stayner LR, Cummings J, Andersen J, Jobe CM. Shoulder dislocations in patients older than 40 years of age. Orthop Clin North Am. 2000 Apr;31(2):231-9. doi: 10.1016/s0030-5898(05)70143-7. PMID 10736392
- [Background] Shin SJ, Yun YH, Kim DJ, Yoo JD. Treatment of traumatic anterior shoulder dislocation in patients older than 60 years. Am J Sports Med. 2012 Apr;40(4):822-7. doi: 10.1177/0363546511434522. Epub 2012 Jan 27. PMID 22287643